CLINICAL TRIAL: NCT06649760
Title: Effect of Message Framing Through M-Health on Oral Health Conditions and Oral Health Related Quality of Life Among Refugees in Alexandria, Egypt: A Randomized Controlled Clinical Trial
Brief Title: Oral Health Education and Message Framing Effect on Oral Health Status of Refugees in Egypt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Dina Youssef Attia, Assistant lecturer, Dr., Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Refugees oral health education
Record Dates: First submitted 2024-10-12; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Knowledge, Attitudes, Practice; Caries,Dental; Plaque, Dental; Gingivitis; Pocket, Periodontal
Keywords: Dental caries; Plaque; KAP; Gingivitis
MeSH Terms: conditions — Behavior; Dental Caries; Dental Plaque; Gingivitis; Periodontal Pocket; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gain-framed messages (Experimental): The participants will receive every 2 weeks a boosting reminder mobile text message in a gain-framed way. For example, "Great breath, healthy gums only a toothbrush away" "flossing your teeth daily removes particles of food in the mouth, avoiding bacteria, which promotes great breath."
  Interventions: Behavioral: Gain and loss framed mobile text messages
- Loss-framed message (Experimental): he participants will receive every 2 weeks a boosting reminder mobile text message in a loss-framed way. For example, "Brush now and avoid bad breath and gum disease", "If you don't floss your teeth daily, particles of food remain in the mouth, collecting bacteria, which causes bad breath."
  Interventions: Behavioral: Gain and loss framed mobile text messages
- Control group (No Intervention): Participants allocated to this group will not receive mobile text messages. They will only receive the oral health education session given to all participants at the beginning.

INTERVENTIONS:
Behavioral: Gain and loss framed mobile text messages — To assess the effect of message framing on enhancing oral health practices in a group of refugees
  Arms: Gain-framed messages; Loss-framed message

SUMMARY:
Refugees, facing forced displacement and often exposed to traumatic experiences, represent a vulnerable population with unique healthcare needs. Oral health is considered a prominent factor that contributes to quality of life.

Therefore, this study aim at assessing the effect of message framing on enhancing oral health practices in a group of refugees in Alexandria, Egypt. A three-arm cluster randomized controlled clinical trial will compare a gain-framed mobile text messages group, a loss-framed mobile text messages group, and a control group. The primary outcome is the improvement in oral health practices measured by changes in dental plaque and secondary outcome is to assess change in oral health-related quality of life. In addition, oral health knowledge, attitudes, and practices of refugees will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Refugees older than 18 years old.
* From Arabic speaking countries.
* Has been resident in Alexandria, Egypt for at least 6 months.
* Having mobile phones to receive text messages.
* Agrees to participate in the study.

Exclusion Criteria:

* Planning to move away during 1 year study period.
* Participating in any kind of oral health education and promotion programs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-06-29 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Oral health knowledge improvement | Immediately after structured oral health session, 6 months and 1 year after baseline
  To assess change in level of oral health knowledge before and after program using a validated questionnaire
Oral health practices improvement | 6 months and 1 year after baseline
  Assess toothbrushing and flossing frequency before and after the education session and reminder mobile messages
Oral hygiene status assesment | 6 months and 1 year after baseline
  measure the change in plaque index scores among participants
Gingival health assessment | 6 months and 1 year after baseline
  measure the change in gingival index scores among participants
Periodontal health status | 6 months and 1 year after baseline
  measure the change in CPI index scores among participants

CONTACTS AND LOCATIONS:
Overall Officials: Mona El Kashlan, Professor, Study Director — Alexandria University
Locations (1):
- Caritas, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
Study protocol and assessment forms.